CLINICAL TRIAL: NCT01698918
Title: An Open-label, Phase II, Single-arm Study of Everolimus in Combination With Letrozole in the Treatment of Postmenopausal Women With Estrogen Receptor Positive HER2 Negative Metastatic or Locally Advanced Breast Cancer
Brief Title: Open-label, Phase II, Study of Everolimus Plus Letrozole in Postmenopausal Women With ER+, HER2- Metastatic or Locally Advanced Breast Cancer
Acronym: BOLERO-4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001Y24135; 2012-003065-17 (EudraCT Number)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Hormone Receptor Positive Breast Cancer
Keywords: Metastatic breast cancer; Locally advanced breast cancer; HER2-; ER+; Everolimus; Afinitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Everolimus; Letrozole; exemestane; Ethanol

STUDY DESIGN:
Intervention Model Description: The main study was an open-label single-arm study. The stomatitis sub-study was a randomized open-label study with two arms: dexamethasone and standard of care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Everolimus+letrozole/exemestane (first line and second line treatment) (Experimental): Participants received everolimus in combination with letrozole as first-line treatment. Only participants who had disease progression in the first line setting (core phase) were offered second-line treatment (everolimus in combination with exemestane)
  Interventions: Drug: Everolimus; Drug: Letrozole; Drug: Exemestane; Drug: Alcohol-free dexamethasone mouth rinse (Stomatitis sub-study); Drug: Standard of care to treat stomatitis (Stomatitis sub-study)

INTERVENTIONS:
Drug: Everolimus — Everolimus was self-administered as a daily dose of 10mg (two 5mg tablets) taken orally continuously until progression of disease, unacceptable toxicity or withdrawal of consent.
  Other Names: RAD001
Drug: Letrozole — 1st line study treatment: Letrozole was self administered as a daily dose of 2.5mg continuously until disease progression or any other reason for which the patient might be discontinued
  Other Names: Femara
Drug: Exemestane — 2nd Line Study Treatment: Exemestane was self administered as a daily dose of 25mg taken orally continuously until disease progression or any other reason for which the patient might be discontinued
  Other Names: Aromasin
Drug: Alcohol-free dexamethasone mouth rinse (Stomatitis sub-study) — Alcohol-free 0.5mg/5ml dexamethasone oral solution was self-administered at a daily dose of 10ml 3 times per day (participants with confirmed stomatitis who entered the stomatitis sub-study).
Drug: Standard of care to treat stomatitis (Stomatitis sub-study) — Standard of care used to treat stomatitis at the patient's center (participants with confirmed stomatitis who entered the stomatitis sub-study).

SUMMARY:
The purpose of this study was to assess the efficacy and safety of first-line treatment with everolimus plus letrozole in postmenopausal women with estrogen receptor-positive (ER+), human epidermal growth factor receptor 2 negative (HER2-) locally advanced or metastatic breast cancer.

Moreover, the study also aimed to investigate the efficacy and safety of second line treatment with everolumus plus examestane in participants whose disease progressed during everolimus plus letrozole therapy.

DETAILED DESCRIPTION:
This was an open-label, phase II, multicenter, international, single-arm study for postmenopausal women with ER+/HER2- metastatic or locally advanced breast cancer.

This study was comprised of 2 phases:

- Core Phase: from first participant first visit to 24 months after enrollment of the last participant (and upon approval of amendment 5 dated 14-Feb-2017), up to approximately 4 years. The main purpose of the amendment 5 was to implement an Extension Phase up to 3 years.

During the core phase, all enrolled participants received everolimus in combination with letrozole in the first line setting until disease progression or any other reason for which the participant might be discontinued. Only those participants who had disease progression in the first line setting were offered second line treatment (everolimus in combination with exemestane). Participants who discontinued first line treatment due to reasons other than disease progression were not eligible for second line treatment. The participants who were treated in the second line setting continued treatment until disease progression, unacceptable toxicity or withdrawal of consent.

- Extension Phase: Participants that were still benefiting from everolimus at the end of the Core Phase (and upon approval of amendment 5 dated 14-Feb-2017) were transitioned to the Extension phase of the study. Participants were continued on their existing line of treatment (everolimus plus letrozole or everolimus plus exemestane) in the extension, up to 3 years or until progression or any other reason for which the participant might be discontinued. Participants entering the Extension Phase on first line treatment and deemed to no longer be clinically benefiting were not offered second line treatment in the context of the study

This study included a randomized, open-label sub-study for participants in countries where the alcohol-free 0.5mg/5ml dexamethasone oral solution was commercially available who experienced a stomatitis event: at the first onset of symptoms suggestive of stomatitis, participants were to contact the study site and based on preliminary confirmation of diagnosis, participants were asked to visit the study site within 24 hours. Upon confirmation of stomatitis, participants in countries where the alcohol-free 0.5 mg/5 mL dexamethasone oral solution was commercially available (US sites only) were randomly assigned in a 1:1 ratio to take either 0.5 mg/5 mL dexamethasone mouth rinse or the standard of care used to treat stomatitis at the participant's center.

All participants who experienced stomatitis (regardless of inclusion in the sub-study) were instructed to fill out the Oral Stomatitis Daily Questionnaire (OSDQ) at home every day until the participant recovered. For subsequent episodes of stomatitis, participants were instructed to contact the physician. If part of the randomized set upon telephone confirmation, they were instructed to utilize the same treatment they were assigned to after the first episode and complete the OSDQ booklet.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic or locally advanced, unresectable breast cancer not amenable to curative treatment by surgery or radiotherapy
* Histological or cytological confirmation of ER+/ HER2- breast cancer
* Postmenopausal women
* No prior treatment for metastatic breast cancer

Exclusion Criteria:

* Patients with only non-measurable lesions other than bone metastases (e.g., pleural effusion, ascites, etc)
* Patients who had received prior hormonal or any other systemic therapy for metastatic breast cancer. Patients might have received prior neoadjuvant or adjuvant endocrine therapy. In the case of neoadjuvant or adjuvant NSAI (letrozole/anastrozole) therapy patients must have completed therapy at least 1 year prior to study enrollment.
* Previous treatment with mTOR inhibitors.
* Known hypersensitivity to mTOR inhibitors, e.g., sirolimus (rapamycin).

Other protocol-defined inclusion/exclusion criteria might apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-03-07 (Actual); Primary Completion 2015-12-17 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (46):
- United States (15):
  - University of Alabama Comprehensive Cancer Center SC-2, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Loma Linda University Loma Linda, Loma Linda, California
  - Breastlink Medical Group Dept. of BreastlinkResearchGrp, Long Beach, California
  - Oncology Specialists, SC Advocate Medical Group-Niles, Park Ridge, Illinois
  - St. Francis Health Comprehensive Cancer Center, Topeka, Kansas
  - Norton Healthcare Inc SC, Louisville, Kentucky
  - Baystate Medical Center SC-2, Springfield, Massachusetts
  - Saint Barnabas Medical Center CancerCenter of Saint Barnabas, Livingston, New Jersey
  - University of New Mexico Hospital SC, Albuquerque, New Mexico
  - Broome Oncology SC, Johnson City, New York
  - Columbia University Medical Center- New York Presbyterian Columbia, New York, New York
  - Cone Health Cancer Center, Greensboro, North Carolina
  - East Texas Hematology Clinic SC, Lufkin, Texas
  - Utah Cancer Specialists Dept.of Utah Cancer Spec. (3), Salt Lake City, Utah
- Argentina (2):
  - Novartis Investigative Site, Santa Rosa, La Pampa Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
- Brazil (2):
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- France (7):
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Hyères
  - Novartis Investigative Site, Le Chesnay
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nancy
  - Novartis Investigative Site, Nantes
- Hungary (3):
  - Novartis Investigative Site, Kecskemét, Bács-Kiskun county
  - Novartis Investigative Site, Gyula
  - Novartis Investigative Site, Szekszárd
- Japan (5):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Shiwa-gun, Iwate
  - Novartis Investigative Site, Kawasaki, Kanagawa
  - Novartis Investigative Site, Kumamoto, Kumamoto
- Novartis Investigative Site, Maastricht, AZ, Netherlands
- Portugal (2):
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Porto
- Novartis Investigative Site, Seoul, South Korea
- Spain (3):
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Antalya
  - Novartis Investigative Site, Istanbul
  - Novartis Investigative Site, Izmir
- Novartis Investigative Site, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Royce M, Bachelot T, Villanueva C, Ozguroglu M, Azevedo SJ, Cruz FM, Debled M, Hegg R, Toyama T, Falkson C, Jeong J, Srimuninnimit V, Gradishar WJ, Arce C, Ridolfi A, Lin C, Cardoso F. Everolimus Plus Endocrine Therapy for Postmenopausal Women With Estrogen Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative Advanced Breast Cancer: A Clinical Trial. JAMA Oncol. 2018 Jul 1;4(7):977-984. doi: 10.1001/jamaoncol.2018.0060. PMID 29566104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 52 centers in 13 countries.
Pre-assignment Details: A total of 245 participants were screened of which 202 participants were enrolled in this study to receive study treatment.
Groups:
- Everolimus+Letrozole/Exemestane (First-line Treatment and Second-line Treatment): Participants received everolimus in combination with letrozole as first line treatment. Only participants who had disease progression in the first line setting (core phase) were offered second-line treatment (everolimus in combination with exemestane)
Period: First Line Treatment (Core+Extension)
Arm/Group | Everolimus+Letrozole/Exemestane (First-line Treatment and Second-line Treatment)
Started | 202
Dexamethasone Randomized Set (Stomatitis Sub-study) (Participants experiencing stomatitis (in countries where the alcohol-free 0.5 mg/5 mL dexamethasone oral solution was commercially available) randomized to take 0.5 mg/5 mL dexamethasone mouth rinse.) | 11
Standard of Care Randomized Set (Stomatitis Sub-study) (Participants experiencing stomatitis (in countries where the alcohol-free 0.5 mg/5 mL dexamethasone oral solution was commercially available) randomized to take standard of care to treat stomatitis) | 13
Completed | 29
Not Completed | 173
Not completed — Adverse Event | 33
Not completed — Withdrawal by Subject | 11
Not completed — Death | 2
Not completed — Disease progression | 120
Not completed — Physician Decision | 7
Period: Second Line Treatment (Core+Extension)
Arm/Group | Everolimus+Letrozole/Exemestane (First-line Treatment and Second-line Treatment)
Started | 53
Completed | 7
Not Completed | 46
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Death | 1
Not completed — Disease progression | 38
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus+Letrozole/Exemestane (First-line Treatment and Second-line Treatment)
Number analyzed (Participants) | 202
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (8.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 146
  Black | 7
  Asian | 44
  Pacific islander | 1
  Other | 4

OUTCOME MEASURES:

1. Primary Outcome: First-line Treatment: Progression-free Survival (PFS)
Description: PFS in the first line setting is defined as the time from the date of enrollment to the date of first documented progression based on local radiology review or death due to any cause. If a participant did not progress or was not known to have died at the date of the analysis cut-off or start of another antineoplastic therapy, the PFS date was censored to the date of last adequate tumor assessment prior to cut-off date or start of antineoplastic therapy. The median PFS was estimated and presented along with 95% confidence intervals. The primary analysis of PFS for first line was performed 12 months after the last patient's recruitment.
Time Frame: From the date of enrollment to the date of first documented progression or deaths, assessed up to approximately 2.8 years
Population: Full Analysis Set (FAS): All participants to whom the first-line study treatment was assigned
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Everolimus+Letrozole (First-line Treatment): Participants received everolimus in combination with letrozole as first-line treatment.
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 202
Months | NA [18.0 to NA] — Not applicable (NA) indicates median PFS was not reached

2. Secondary Outcome: First-line Treatment: Overall Response Rate (ORR)
Description: ORR in first line setting is defined as the percentage of participants while on first-line treatment with best overall response of complete response (CR) or partial response (PR) according to RECIST version 1.0 based on local review. Confidence intervals were calculated based on the Exact Clopper-Pearson method.
  ORR while on first-line treatment was assessed up to 24 months after the last patient's recruitment.
  CR: disappearance of all target lesions PR: at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
Time Frame: From the date of enrollment until discontinuation of first-line treatment, assessed up to approximately 3.8 years
Population: FAS: All participants to whom the first-line study treatment was assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Everolimus+Letrozole (First Line Treatment): Participants received everolimus in combination with letrozole as first-line treatment
Arm/Group | Everolimus+Letrozole (First Line Treatment)
Number analyzed (Participants) | 202
Percentage of participants | 45.0 [38.1 to 52.2]

3. Secondary Outcome: First-line Treatment: Clinical Benefit Rate (CBR)
Description: CBR in first line is defined as the percentage of participants while on first-line treatment with best overall response of CR, PR or stable disease (SD) with a duration of 24 weeks or longer, according to RECIST version 1.0 based on local review. Confidence intervals (CI) were calculated based on the Exact Clopper-Pearson method.
  CBR while on first-line treatment was assessed up to 24 months after the last patient's recruitment.
  CR: disappearance of all target lesions PR: at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease
Time Frame: From the date of enrollment until first-line treatment discontinuation, assessed up to approximately 3.8 years
Population: FAS: All participants to whom the first-line study treatment was assigned
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 202
Percentage of participants | 74.3 [67.7 to 80.1]

4. Secondary Outcome: Second-line Treatment: Progression-free Survival (PFS)
Description: PFS in the second line setting is defined as the time interval between the start of the second-line treatment and documented disease progression based on local radiology review or death due to any cause reported during or after second-line treatment period. If a participant did not progress or was not known to have died at the date of the analysis cut-off or start of another antineoplastic therapy, the PFS date was censored to the date of last adequate tumor assessment prior to cut-off date or start of antineoplastic therapy. The median PFS was estimated and presented along with 95% confidence intervals.
  PFS while on second-line treatment was assessed up to 24 months after the last patient's recruitment.
Time Frame: From the start of the second-line treatment until the date of first documented progression or death, assessed up to approximately 2.4 years
Population: Participants in the Full Analysis Set second line (FAS-2L), including all participants in the FAS who received at least one dose of second-line study medication, with evaluable data for this endpoint.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Everolimus+Exemestane (Second Line Treatment): Participants who had disease progression in the first line setting (core phase) were treated with second line treatment (everolimus in combination with exemestane)
Arm/Group | Everolimus+Exemestane (Second Line Treatment)
Number analyzed (Participants) | 50
Months | 3.7 [1.9 to 7.4]

5. Secondary Outcome: Second-line Treatment: Overall Response Rate (ORR)
Description: ORR in second line is defined as the percentage of participants receiving second-line study treatment with best overall response of complete response (CR) or partial response (PR) according to RECIST version 1.0 based on local review. Confidence intervals (CI) were calculated based on the Exact Clopper-Pearson method.
  ORR while on second-line treatment was assessed up to 24 months after the last patient's recruitment.
  CR: disappearance of all target lesions PR: at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters
Time Frame: From the start of the second-line treatment up to approximately 2.4 years
Population: Participants in the FAS-2L, including all participants in the FAS who received at least one dose of second-line study medication, with evaluable data for this endpoint
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Everolimus+Exemestane (Second-line Treatment): Participants who had disease progression in the first line setting (core phase) were treated with second-line treatment (everolimus in combination with exemestane)
Arm/Group | Everolimus+Exemestane (Second-line Treatment)
Number analyzed (Participants) | 50
Percentage of participants | 6.0 [1.3 to 16.5]

6. Secondary Outcome: Second-line Treatment: Clinical Benefit Rate (CBR)
Description: CBR in second line is defined as the percentage of participants receiving second-line study treatment with best overall response of CR, PR or stable disease (SD) with a duration of 24 weeks or longer, according to RECIST version 1.0 based on local review. Confidence intervals (CI) were calculated based on the Exact Clopper-Pearson method.
  CBR while on second-line treatment was assessed up to 24 months after the last patient's recruitment.
  CR: disappearance of all target lesions PR: at least a 30% decrease in the sum of the longest diameter of all target lesions, taking as reference the baseline sum of the longest diameters.
  SD: Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for progressive disease
Time Frame: From the start of the second-line treatment up to approximately 2.4 years
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Everolimus+Exemestane (Second-line Treatment)
Number analyzed (Participants) | 50
Percentage of participants | 28.0 [16.2 to 42.5]

7. Secondary Outcome: Overall Survival (OS)
Description: OS following first-line treatment with everolimus + letrozole is defined as the time from the date of receiving first line study treatment to date of death due to any cause (including first-line and second-line treatment periods). If a participant was not known to have died, survival was censored at the date of last contact.
  OS following first-line treatment was assessed up to 24 months after last patient's recruitment.
Time Frame: From the date of enrollment to date of death, assessed up to approximately 3.8 years
Population: FAS: All participants to whom the first-line study treatment was assigned
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Everolimus+Letrozole/Exemestane (First-line Treatment and Second-line Treatment)
Number analyzed (Participants) | 202
Months | NA [37.0 to NA] — Not applicable (NA) indicates median OS was not reached

8. Secondary Outcome: First-line Treatment: Time to First Stomatitis Episode as Assessed by the Oral Stomatitis Daily Questionnaire (OSDQ)
Description: The time to first occurrence of stomatitis based on OSDQ is defined as time from first-line treatment administration to start date of the stomatitis episode recorded in the OSDQ in the first line. The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The first item asked the participants when they experienced the first symptoms of stomatitis. Start date of the first occurrence of stomatitis is defined as the first date ever recorded for this item in the questionnaire. Patient reported outcomes (PROs) were assessed up to 24 months after last patient's recruitment.
Time Frame: From first-line treatment administration until first stomatitis episode in the first line, assessed up to approximately 3.8 years
Population: First-line stomatitis analysis set (SAS-1L): All participants in the FAS who agreed to fill in the OSDQ and who developed their first stomatitis event (based on OSDQ) in the first line.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 92
Weeks | 1.7 [1.3 to 2.1]

9. Secondary Outcome: First-line Treatment: Duration of First Stomatitis Based on OSDQ
Description: The duration of the first stomatitis episode was calculated using the start and end date recorded in the OSDQ. The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis. The first item of the questionnaire asked the participants the date when they experienced the first symptoms of stomatitis. Start date of the first occurrence of stomatitis is defined as the first date ever recorded for this item in the questionnaire. Stop date of the first stomatitis episode is defined as the last date the OSDQ was completed for this episode. Participants were censored if they died before resolution of stomatitis, received a new anticancer therapy, discontinued the study treatment with no resolution of the stomatitis or the stomatitis event was still on-going at the cut-off. PROs were assessed up to 24 months after last patient's recruitment.
Time Frame: From start date of first stomatitis episode in first line until its resolution, assessed up to 3.8 years
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 92
Weeks | 12.3 [4.1 to 23.1]

10. Secondary Outcome: First-line Treatment: Number of Participants With Shift of Response in OSDQ Score on Overall Health at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily up to the resolution of the stomatitis episode. The second item asked the participant to rate their overall health from 0 (worst possible) to 10 (perfect health). The overall health OSDQ scores are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 92
Participants
  From 0 (Day 1) to 0 (end of first stomatitis) | 2
  From 0 (Day 1) to 1 (end of first stomatitis) | 1
  From 0 (Day 1) to 5 (end of first stomatitis) | 1
  From 1 (Day 1) to 1 (end of first stomatitis) | 1
  From 1 (Day 1) to 2 (end of first stomatitis) | 1
  From 2 (Day 1) to 5 (end of first stomatitis) | 1
  From 2 (Day 1) to 8 (end of first stomatitis) | 2
  From 3 (Day 1) to 0 (end of first stomatitis) | 1
  From 3 (Day 1) to 3 (end of first stomatitis) | 3
  From 3 (Day 1) to 5 (end of first stomatitis) | 2
  From 3 (Day 1) to 10 (end of first stomatitis) | 2
  From 4 (Day 1) to 3 (end of first stomatitis) | 2
  From 4 (Day 1) to 5 (end of first stomatitis) | 1
  From 4 (Day 1) to 7 (end of first stomatitis) | 1
  From 4 (Day 1) to 8 (end of first stomatitis) | 2
  From 5 (Day 1) to 0 (end of first stomatitis) | 1
  From 5 (Day 1) to 3 (end of first stomatitis) | 3
  From 5 (Day 1) to 4 (end of first stomatitis) | 1
  From 5 (Day 1) to 5 (end of first stomatitis) | 7
  From 5 (Day 1) to 6 (end of first stomatitis) | 4
  From 5 (Day 1) to 7 (end of first stomatitis) | 3
  From 5 (Day 1) to 9 (end of first stomatitis) | 1
  From 5 (Day 1) to 10 (end of first stomatitis) | 2
  From 6 (Day 1) to 5 (end of first stomatitis) | 2
  From 6 (Day 1) to 6 (end of first stomatitis) | 3
  From 6 (Day 1) to 7 (end of first stomatitis) | 2
  From 6 (Day 1) to 9 (end of first stomatitis) | 2
  From 7 (Day 1) to 3 (end of first stomatitis) | 2
  From 7 (Day 1) to 4 (end of first stomatitis) | 1
  From 7 (Day 1) to 5 (end of first stomatitis) | 1
  From 7 (Day 1) to 7 (end of first stomatitis) | 3
  From 7 (Day 1) to 9 (end of first stomatitis) | 1
  From 8 (Day 1) to 1 (end of first stomatitis) | 1
  From 8 (Day 1) to 7 (end of first stomatitis) | 1
  From 8 (Day 1) to 8 (end of first stomatitis) | 4
  From 8 (Day 1) to 9 (end of first stomatitis) | 5
  From 8 (Day 1) to 10 (end of first stomatitis) | 2
  From 9 (Day 1) to 0 (end of first stomatitis) | 1
  From 9 (Day 1) to 4 (end of first stomatitis) | 2
  From 9 (Day 1) to 8 (end of first stomatitis) | 1
  From 9 (Day 1) to 9 (end of first stomatitis) | 8
  From 10 (Day 1) to 3 (end of first stomatitis) | 1
  From 10 (Day 1) to 9 (end of first stomatitis) | 1
  From missing value (Day 1) to missing value (end of first stomatitis) | 3

11. Secondary Outcome: First-line Treatment: Number of Participants With Shift of Response in OSDQ Score on Mouth and Throat Soreness at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The third item asked the participant to rate their mouth and throat soreness from 0 (no soreness) to 4 (extreme soreness). The mouth and throat soreness OSDQ scores are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 92
Participants
  From 0 (Day 1) to 0 (end of first stomatitis) | 3
  From 1 (Day 1) to 0 (end of first stomatitis) | 22
  From 1 (Day 1) to 1 (end of first stomatitis) | 12
  From 1 (Day 1) to 2 (end of first stomatitis) | 3
  From 2 (Day 1) to 0 (end of first stomatitis) | 13
  From 2 (Day 1) to 1 (end of first stomatitis) | 7
  From 2 (Day 1) to 2 (end of first stomatitis) | 4
  From 2 (Day 1) to 3 (end of first stomatitis) | 1
  From 3 (Day 1) to 0 (end of first stomatitis) | 9
  From 3 (Day 1) to 1 (end of first stomatitis) | 4
  From 3 (Day 1) to 2 (end of first stomatitis) | 5
  From 3 (Day 1) to 3 (end of first stomatitis) | 1
  From 3 (Day 1) to 4 (end of first stomatitis) | 1
  From 4 (Day 1) to 1 (end of first stomatitis) | 2
  From 4 (Day 1) to 2 (end of first stomatitis) | 1
  From missing value (Day 1) to missing value (end of first stomatitis) | 4

12. Secondary Outcome: First-line Treatment: Number of Participants With Shift of Response in OSDQ Score on Mouth and Throat Soreness Limiting Swallowing, Drinking, Eating, Talking and Sleeping at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The fourth item asked the participant to rate how much their mouth and throat soreness limited them in 1) swallowing, 2) drinking, 3) eating, 4) talking and 5) sleeping. For each activity, mouth and throat soreness scores ranged from 0 (not limited) to 4 (unable to do). Scores are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First Line Treatment)
Number analyzed (Participants) | 92
Participants
  Swallowing: From 0 (Day 1) to 0 (end of first stomatitis) | 40
  Swallowing: From 0 (Day 1) to 1 (end of first stomatitis) | 3
  Swallowing: From 0 (Day 1) to 2 (end of first stomatitis) | 1
  Swallowing: From 1 (Day 1) to 0 (end of first stomatitis) | 7
  Swallowing: From 1 (Day 1) to 1 (end of first stomatitis) | 6
  Swallowing: From 1 (Day 1) to 2 (end of first stomatitis) | 3
  Swallowing: From 1 (Day 1) to 3 (end of first stomatitis) | 1
  Swallowing: From 2 (Day 1) to 0 (end of first stomatitis) | 6
  Swallowing: From 2 (Day 1) to 1 (end of first stomatitis) | 4
  Swallowing: From 2 (Day 1) to 2 (end of first stomatitis) | 2
  Swallowing: From 3 (Day 1) to 0 (end of first stomatitis) | 8
  Swallowing: From 3 (Day 1) to 1 (end of first stomatitis) | 2
  Swallowing: From 3 (Day 1) to 3 (end of first stomatitis) | 2
  Swallowing: From missing value (Day 1) to missing value (end of first stomatitis) | 7
  Drinking: From 0 (Day 1) to 0 (end of first stomatitis) | 48
  Drinking: From 0 (Day 1) to 1 (end of first stomatitis) | 4
  Drinking: From 0 (Day 1) to 2 (end of first stomatitis) | 1
  Drinking: From 1 (Day 1) to 0 (end of first stomatitis) | 10
  Drinking: From 1 (Day 1) to 1 (end of first stomatitis) | 5
  Drinking: From 1 (Day 1) to 2 (end of first stomatitis) | 1
  Drinking: From 2 (Day 1) to 0 (end of first stomatitis) | 4
  Drinking: From 2 (Day 1) to 1 (end of first stomatitis) | 3
  Drinking: From 2 (Day 1) to 2 (end of first stomatitis) | 3
  Drinking: From 2 (Day 1) to 3 (end of first stomatitis) | 2
  Drinking: From 3 (Day 1) to 0 (end of first stomatitis) | 6
  Drinking: From 3 (Day 1) to 1 (end of first stomatitis) | 1
  Drinking: From 3 (Day 1) to 3 (end of first stomatitis) | 1
  Drinking: From missing value (Day 1) to missing value (end of first stomatitis) | 9
  Eating: From 0 (Day 1) to 0 (end of first stomatitis) | 17
  Eating: From 0 (Day 1) to 1 (end of first stomatitis) | 2
  Eating: From 0 (Day 1) to 2 (end of first stomatitis) | 1
  Eating: From 1 (Day 1) to 0 (end of first stomatitis) | 14
  Eating: From 1 (Day 1) to 1 (end of first stomatitis) | 11
  Eating: From 1 (Day 1) to 2 (end of first stomatitis) | 2
  Eating: From 2 (Day 1) to 0 (end of first stomatitis) | 8
  Eating: From 2 (Day 1) to 1 (end of first stomatitis) | 3
  Eating: From 2 (Day 1) to 2 (end of first stomatitis) | 4
  Eating: From 2 (Day 1) to 3 (end of first stomatitis) | 2
  Eating: From 3 (Day 1) to 0 (end of first stomatitis) | 7
  Eating: From 3 (Day 1) to 1 (end of first stomatitis) | 6
  Eating: From 3 (Day 1) to 2 (end of first stomatitis) | 3
  Eating: From 3 (Day 1) to 3 (end of first stomatitis) | 4
  Eating: From 4 (Day 1) to 1 (end of first stomatitis) | 1
  Eating: From missing value (Day 1) to missing value (end of first stomatitis) | 7
  Talking: From 0 (Day 1) to 0 (end of first stomatitis) | 45
  Talking: From 0 (Day 1) to 1 (end of first stomatitis) | 5
  Talking: From 1 (Day 1) to 0 (end of first stomatitis) | 12
  Talking: From 1 (Day 1) to 1 (end of first stomatitis) | 2
  Talking: From 2 (Day 1) to 0 (end of first stomatitis) | 5
  Talking: From 2 (Day 1) to 1 (end of first stomatitis) | 2
  Talking: From 2 (Day 1) to 2 (end of first stomatitis) | 3
  Talking: From 2 (Day 1) to 3 (end of first stomatitis) | 1
  Talking: From 3 (Day 1) to 0 (end of first stomatitis) | 4
  Talking: From 3 (Day 1) to 2 (end of first stomatitis) | 1
  Talking: From 3 (Day 1) to 3 (end of first stomatitis) | 3
  Talking: From missing value (Day 1) to missing value (end of first stomatitis) | 9
  Sleeping: From 0 (Day 1) to 0 (end of first stomatitis) | 48
  Sleeping: From 0 (Day 1) to 1 (end of first stomatitis) | 4
  Sleeping: From 0 (Day 1) to 2 (end of first stomatitis) | 1
  Sleeping: From 1 (Day 1) to 0 (end of first stomatitis) | 8
  Sleeping: From 1 (Day 1) to 1 (end of first stomatitis) | 2
  Sleeping: From 1 (Day 1) to 2 (end of first stomatitis) | 2
  Sleeping: From 2 (Day 1) to 0 (end of first stomatitis) | 4
  Sleeping: From 2 (Day 1) to 1 (end of first stomatitis) | 3
  Sleeping: From 2 (Day 1) to 2 (end of first stomatitis) | 6
  Sleeping: From 3 (Day 1) to 0 (end of first stomatitis) | 1
  Sleeping: From 3 (Day 1) to 1 (end of first stomatitis) | 1
  Sleeping: From 3 (Day 1) to 2 (end of first stomatitis) | 1
  Sleeping: From missing value (Day 1) to missing value (end of first stomatitis) | 11

13. Secondary Outcome: First-line Treatment: Number of Participants With Shift of Response in OSDQ Score on Mouth Pain Severity at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The fifth item asked the participant to rate their mouth pain severity from 0 (no pain) to 10 (unbearable pain). The mouth pain severity OSDQ scores are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 92
Participants
  From 0 (Day 1) to 0 (end of first stomatitis) | 5
  From 1 (Day 1) to 0 (end of first stomatitis) | 10
  From 1 (Day 1) to 1 (end of first stomatitis) | 6
  From 1 (Day 1) to 2 (end of first stomatitis) | 1
  From 1 (Day 1) to 3 (end of first stomatitis) | 1
  From 1 (Day 1) to 5 (end of first stomatitis) | 1
  From 2 (Day 1) to 0 (end of first stomatitis) | 6
  From 2 (Day 1) to 3 (end of first stomatitis) | 1
  From 3 (Day 1) to 0 (end of first stomatitis) | 7
  From 3 (Day 1) to 1 (end of first stomatitis) | 1
  From 3 (Day 1) to 2 (end of first stomatitis) | 2
  From 3 (Day 1) to 3 (end of first stomatitis) | 1
  From 3 (Day 1) to 4 (end of first stomatitis) | 2
  From 4 (Day 1) to 0 (end of first stomatitis) | 4
  From 4 (Day 1) to 1 (end of first stomatitis) | 2
  From 4 (Day 1) to 4 (end of first stomatitis) | 1
  From 4 (Day 1) to 5 (end of first stomatitis) | 1
  From 5 (Day 1) to 0 (end of first stomatitis) | 3
  From 5 (Day 1) to 1 (end of first stomatitis) | 1
  From 5 (Day 1) to 2 (end of first stomatitis) | 1
  From 5 (Day 1) to 3 (end of first stomatitis) | 1
  From 5 (Day 1) to 4 (end of first stomatitis) | 1
  From 5 (Day 1) to 5 (end of first stomatitis) | 1
  From 5 (Day 1) to 6 (end of first stomatitis) | 1
  From 5 (Day 1) to 7 (end of first stomatitis) | 1
  From 5 (Day 1) to 10 (end of first stomatitis) | 1
  From 6 (Day 1) to 0 (end of first stomatitis) | 2
  From 6 (Day 1) to 1 (end of first stomatitis) | 1
  From 6 (Day 1) to 2 (end of first stomatitis) | 1
  From 6 (Day 1) to 5 (end of first stomatitis) | 1
  From 6 (Day 1) to 6 (end of first stomatitis) | 1
  From 6 (Day 1) to 8 (end of first stomatitis) | 1
  From 7 (Day 1) to 0 (end of first stomatitis) | 2
  From 7 (Day 1) to 1 (end of first stomatitis) | 2
  From 7 (Day 1) to 2 (end of first stomatitis) | 1
  From 7 (Day 1) to 7 (end of first stomatitis) | 1
  From 8 (Day 1) to 0 (end of first stomatitis) | 3
  From 8 (Day 1) to 2 (end of first stomatitis) | 1
  From 8 (Day 1) to 4 (end of first stomatitis) | 2
  From 8 (Day 1) to 5 (end of first stomatitis) | 1
  From 8 (Day 1) to 6 (end of first stomatitis) | 1
  From 8 (Day 1) to 9 (end of first stomatitis) | 1
  From 9 (Day 1) to 0 (end of first stomatitis) | 2
  From 9 (Day 1) to 9 (end of first stomatitis) | 1
  From missing value (Day 1) to missing value (end of first stomatitis) | 4

14. Secondary Outcome: First-line Treatment: Number of Participants With Shift of Response in OSDQ Score on Mouth Pain Severity Affecting Daily Activities at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The sixth item asked the participant to rate their mouth pain severity affecting daily activities score from 0 (no effect on daily activities) to 10 (completely prevented from doing daily activities). The mouth pain severity affecting daily activities OSDQ scores are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 92
Participants
  From 0 (Day 1) to 0 (end of first stomatitis) | 33
  From 0 (Day 1) to 1 (end of first stomatitis) | 1
  From 0 (Day 1) to 5 (end of first stomatitis) | 1
  From 1 (Day 1) to 0 (end of first stomatitis) | 7
  From 1 (Day 1) to 1 (end of first stomatitis) | 4
  From 1 (Day 1) to 4 (end of first stomatitis) | 2
  From 2 (Day 1) to 0 (end of first stomatitis) | 6
  From 2 (Day 1) to 1 (end of first stomatitis) | 1
  From 2 (Day 1) to 2 (end of first stomatitis) | 3
  From 2 (Day 1) to 3 (end of first stomatitis) | 1
  From 2 (Day 1) to 4 (end of first stomatitis) | 1
  From 3 (Day 1) to 0 (end of first stomatitis) | 3
  From 3 (Day 1) to 1 (end of first stomatitis) | 3
  From 3 (Day 1) to 2 (end of first stomatitis) | 1
  From 3 (Day 1) to 3 (end of first stomatitis) | 1
  From 3 (Day 1) to 4 (end of first stomatitis) | 1
  From 4 (Day 1) to 0 (end of first stomatitis) | 2
  From 5 (Day 1) to 0 (end of first stomatitis) | 2
  From 5 (Day 1) to 1 (end of first stomatitis) | 1
  From 5 (Day 1) to 2 (end of first stomatitis) | 1
  From 5 (Day 1) to 3 (end of first stomatitis) | 1
  From 5 (Day 1) to 5 (end of first stomatitis) | 1
  From 5 (Day 1) to 6 (end of first stomatitis) | 1
  From 6 (Day 1) to 1 (end of first stomatitis) | 1
  From 6 (Day 1) to 5 (end of first stomatitis) | 1
  From 6 (Day 1) to 8 (end of first stomatitis) | 1
  From 7 (Day 1) to 0 (end of first stomatitis) | 1
  From 8 (Day 1) to 0 (end of first stomatitis) | 1
  From 8 (Day 1) to 8 (end of first stomatitis) | 1
  From 8 (Day 1) to 10 (end of first stomatitis) | 1
  From 9 (Day 1) to 0 (end of first stomatitis) | 1
  From 9 (Day 1) to 8 (end of first stomatitis) | 1
  From 10 (Day 1) to 10 (end of first stomatitis) | 1
  From missing value (Day 1) to missing value (end of first stomatitis) | 4

15. Secondary Outcome: First-line Treatment (Stomatitis Sub-study): Time to First Stomatitis Episode as Assessed by the OSDQ
Description: The time to first occurrence of stomatitis based on OSDQ is defined as time from first study treatment administration in the first line to start date of the first stomatitis episode recorded in the OSDQ. The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The first item asked the participants when they experienced the first symptoms of stomatitis. Start date of the first occurrence of stomatitis is defined as the first date ever recorded for this item in the questionnaire. PROs were assessed up to 24 months after last patient's recruitment.
  Only participants who were randomized in the stomatitis sub-study were included in this analysis.
Time Frame: From first study treatment administration in the first line until first stomatitis episode, assessed up to approximately 3.8 years
Population: Stomatitis randomized set: All participants in the FAS who were randomized in the stomatitis sub-study to receive dexamethasone or standard of care (i.e. participants in countries where the alcohol-free 0.5mg/5ml dexamethasone oral solution was commercially available who experienced a stomatitis event). Number analyzed indicates the number of participants randomized to each intervention
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Everolimus+ Letrozole (First-line Treatment): Participants received everolimus in combination with letrozole as first-line treatment
Arm/Group | Everolimus+ Letrozole (First-line Treatment)
Number analyzed (Participants) | 24
Weeks
  Dexamethasone: number analyzed (Participants) | 11
  Dexamethasone | 1.4 [0.9 to 1.9]
  Standard of care: number analyzed (Participants) | 13
  Standard of care | 2.3 [0.7 to 5.4]

16. Secondary Outcome: First-line Treatment (Stomatitis Sub-study): Duration of First Stomatitis Based on OSDQ
Description: The duration of the first stomatitis was calculated using the start and end date reported in the OSDQ. The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis. The first item asked the participants the date when they experienced the first symptoms of stomatitis. Start date of the first stomatitis is defined as the first date ever recorded for this item in the questionnaire. Stop date of the first stomatitis is defined as the last date the OSDQ was completed for this episode. Participants were censored if they died before resolution of stomatitis, received a new anticancer therapy, discontinued the study treatment with no resolution of the stomatitis or the stomatitis was still on-going at the cut-off. PROs were assessed up to 24 months after last patient's recruitment. Only participants who were randomized in the stomatitis sub-study were included in this analysis.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 24
Weeks
  Dexamethasone: number analyzed (Participants) | 11
  Dexamethasone | NA [NA to NA] — Not Applicable (NA) indicates median duration of stomatitis was non-estimable because only one event was recorded and ten participants were censored
  Standard of Care: number analyzed (Participants) | 13
  Standard of Care | 13.7 [1.4 to 13.7]

17. Secondary Outcome: First-line Treatment (Stomatitis Sub-study): Number of Participants With Shift of Response in OSDQ Score on Overall Health at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The second item asked the participant to rate their overall health from 0 (worst possible) to 10 (perfect health). The overall health OSDQ score are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
  Only participants who were randomized in the stomatitis sub-study were included in this analysis.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 24
Participants
  Dexamethasone: From 2 (Day 1) to 5 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 2 (Day 1) to 5 (end of first stomatitis) | 1
  Dexamethasone: From 4 (Day 1) to 3 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 4 (Day 1) to 3 (end of first stomatitis) | 1
  Dexamethasone: From 5 (Day 1) to 5 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 5 (Day 1) to 5 (end of first stomatitis) | 1
  Dexamethasone: From 5 (Day 1) to 6 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 5 (Day 1) to 6 (end of first stomatitis) | 1
  Dexamethasone: From 5 (Day 1) to 7 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 5 (Day 1) to 7 (end of first stomatitis) | 1
  Dexamethasone: From 6 (Day 1) to 5 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 6 (Day 1) to 5 (end of first stomatitis) | 1
  Dexamethasone: From 6 (Day 1) to 7 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 6 (Day 1) to 7 (end of first stomatitis) | 1
  Dexamethasone: From 7 (Day 1) to 3 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 7 (Day 1) to 3 (end of first stomatitis) | 1
  Dexamethasone: From 8 (Day 1) to 8 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 8 (Day 1) to 8 (end of first stomatitis) | 1
  Dexamethasone: From 8 (Day 1) to 9 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 8 (Day 1) to 9 (end of first stomatitis) | 1
  Dexamethasone: From 9 (Day 1) to 9 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 9 (Day 1) to 9 (end of first stomatitis) | 1
  SoC: From 0 (Day 1) to 5 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 0 (Day 1) to 5 (end of first stomatitis) | 1
  SoC: From 4 (Day 1) to 3 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 4 (Day 1) to 3 (end of first stomatitis) | 1
  SoC: From 4 (Day 1) to 8 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 4 (Day 1) to 8 (end of first stomatitis) | 1
  SoC: From 5 (Day 1) to 5 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 5 (Day 1) to 5 (end of first stomatitis) | 1
  SoC: From 6 (Day 1) to 7 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 6 (Day 1) to 7 (end of first stomatitis) | 1
  SoC: From 7 (Day 1) to 3 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 7 (Day 1) to 3 (end of first stomatitis) | 1
  SoC: From 8 (Day 1) to 9 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 8 (Day 1) to 9 (end of first stomatitis) | 1
  SoC: From 8 (Day 1) to 10 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 8 (Day 1) to 10 (end of first stomatitis) | 1
  SoC: From 9 (Day 1) to 4 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 9 (Day 1) to 4 (end of first stomatitis) | 1
  SoC: From 9 (Day 1) to 9 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 9 (Day 1) to 9 (end of first stomatitis) | 2
  SoC: From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From missing value (Day 1) to missing value (end of first stomatitis) | 2

18. Secondary Outcome: First-line Treatment (Stomatitis Sub-study): Number of Participants With Shift of Response in OSDQ Score on Mouth and Throat Soreness at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The third item asked the participant to rate their mouth and throat soreness from 0 (no soreness) to 4 (extreme soreness). The mouth and throat soreness OSDQ scores are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
  Only participants who were randomized in the stomatitis sub-study were included in this analysis.
Time Frame: From start date of stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 24
Participants
  Dexamethasone: From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 0 (Day 1) to 0 (end of first stomatitis) | 1
  Dexamethasone: From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 1 (Day 1) to 0 (end of first stomatitis) | 3
  Dexamethasone: From 1 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 1 (Day 1) to 1 (end of first stomatitis) | 2
  Dexamethasone: From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 2 (Day 1) to 0 (end of first stomatitis) | 1
  Dexamethasone: From 2 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 2 (Day 1) to 1 (end of first stomatitis) | 3
  Dexamethasone: From 3 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 3 (Day 1) to 1 (end of first stomatitis) | 1
  SoC: From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 1 (Day 1) to 0 (end of first stomatitis) | 1
  SoC: From 1 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 1 (Day 1) to 1 (end of first stomatitis) | 1
  SoC: From 2 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 2 (Day 1) to 1 (end of first stomatitis) | 1
  SoC: From 3 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 3 (Day 1) to 0 (end of first stomatitis) | 2
  SoC: From 3 (Day 1) to 1 (end of first stomatitis: number analyzed (Participants) | 13
  SoC: From 3 (Day 1) to 1 (end of first stomatitis | 1
  SoC: From 3 (Day 1) to 2 (end of first stomatitis: number analyzed (Participants) | 13
  SoC: From 3 (Day 1) to 2 (end of first stomatitis | 3
  SoC: From 4 (Day 1) to 1 (end of first stomatitis: number analyzed (Participants) | 13
  SoC: From 4 (Day 1) to 1 (end of first stomatitis | 1
  SoC: From 4 (Day 1) to 2 (end of first stomatitis: number analyzed (Participants) | 13
  SoC: From 4 (Day 1) to 2 (end of first stomatitis | 1
  SoC: From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From missing value (Day 1) to missing value (end of first stomatitis) | 2

19. Secondary Outcome: First-line Treatment (Stomatitis Sub-study): Number of Participants With Shift of Response in OSDQ Score on Mouth and Throat Soreness Limiting Swallowing, Drinking, Eating, Talking and Sleeping at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The fourth item asked the participant to rate how much their mouth and throat soreness limited them in 1) swallowing, 2) drinking, 3) eating, 4) talking and 5) sleeping. For each activity, mouth and throat soreness scores ranged from 0 (not limited) to 4 (unable to do). Scores are presented as the shift from Day 1 of first stomatitis stomatitis value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first episode value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
  Only participants who were randomized in the stomatitis sub-study were included in this analysis.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 24
Participants
  Swallowing (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Swallowing (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis) | 6
  Swallowing (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Swallowing (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis) | 2
  Swallowing (dexamethasone): From 1 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Swallowing (dexamethasone): From 1 (Day 1) to 1 (end of first stomatitis) | 1
  Swallowing (dexamethasone): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Swallowing (dexamethasone): From 2 (Day 1) to 0 (end of first stomatitis) | 1
  Swallowing (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Swallowing (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis) | 1
  Swallowing (SoC): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Swallowing (SoC): From 0 (Day 1) to 0 (end of first stomatitis) | 5
  Swallowing (SoC): From 1 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 13
  Swallowing (SoC): From 1 (Day 1) to 2 (end of first stomatitis) | 1
  Swallowing (SoC): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Swallowing (SoC): From 2 (Day 1) to 0 (end of first stomatitis) | 1
  Swallowing (SoC): From 2 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Swallowing (SoC): From 2 (Day 1) to 1 (end of first stomatitis) | 2
  Swallowing (SoC): From 3 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Swallowing (SoC): From 3 (Day 1) to 0 (end of first stomatitis) | 1
  Swallowing (SoC): From 3 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Swallowing (SoC): From 3 (Day 1) to 1 (end of first stomatitis) | 1
  Swallowing (SoC): From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  Swallowing (SoC): From missing value (Day 1) to missing value (end of first stomatitis) | 2
  Drinking (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Drinking (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis) | 6
  Drinking (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Drinking (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis) | 2
  Drinking (dexamethasone): From 1 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Drinking (dexamethasone): From 1 (Day 1) to 1 (end of first stomatitis) | 1
  Drinking (dexamethasone): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Drinking (dexamethasone): From 2 (Day 1) to 0 (end of first stomatitis) | 1
  Drinking (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Drinking (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis) | 1
  Drinking (SoC): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Drinking (SoC): From 0 (Day 1) to 0 (end of first stomatitis) | 3
  Drinking (SoC): From 0 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Drinking (SoC): From 0 (Day 1) to 1 (end of first stomatitis) | 2
  Drinking (SoC): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Drinking (SoC): From 2 (Day 1) to 0 (end of first stomatitis) | 3
  Drinking (SoC): From 2 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Drinking (SoC): From 2 (Day 1) to 1 (end of first stomatitis) | 1
  Drinking (SoC): From 3 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Drinking (SoC): From 3 (Day 1) to 0 (end of first stomatitis) | 1
  Drinking (SoC): From 3 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Drinking (SoC): From 3 (Day 1) to 1 (end of first stomatitis) | 1
  Drinking (SoC): From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  Drinking (SoC): From missing value (Day 1) to missing value (end of first stomatitis) | 2
  Eating (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Eating (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis) | 3
  Eating (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Eating (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis) | 1
  Eating (dexamethasone): From 1 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Eating (dexamethasone): From 1 (Day 1) to 1 (end of first stomatitis) | 2
  Eating (dexamethasone): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Eating (dexamethasone): From 2 (Day 1) to 0 (end of first stomatitis) | 1
  Eating (dexamethasone): From 2 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Eating (dexamethasone): From 2 (Day 1) to 1 (end of first stomatitis) | 2
  Eating (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Eating (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis) | 1
  Eating (dexamethasone): From 3 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Eating (dexamethasone): From 3 (Day 1) to 1 (end of first stomatitis) | 1
  Eating (SoC): From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Eating (SoC): From 1 (Day 1) to 0 (end of first stomatitis) | 2
  Eating (SoC): From 1 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Eating (SoC): From 1 (Day 1) to 1 (end of first stomatitis) | 1
  Eating (SoC): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Eating (SoC): From 2 (Day 1) to 0 (end of first stomatitis) | 1
  Eating (SoC): From 3 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Eating (SoC): From 3 (Day 1) to 0 (end of first stomatitis) | 1
  Eating (SoC): From 3 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Eating (SoC): From 3 (Day 1) to 1 (end of first stomatitis) | 2
  Eating (SoC): From 3 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 13
  Eating (SoC): From 3 (Day 1) to 2 (end of first stomatitis) | 3
  Eating (SoC): From 4 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Eating (SoC): From 4 (Day 1) to 1 (end of first stomatitis) | 1
  Eating (SoC): From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  Eating (SoC): From missing value (Day 1) to missing value (end of first stomatitis) | 2
  Talking (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Talking (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis) | 6
  Talking (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Talking (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis) | 1
  Talking (dexamethasone): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Talking (dexamethasone): From 2 (Day 1) to 0 (end of first stomatitis) | 2
  Talking (dexamethasone): From 2 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Talking (dexamethasone): From 2 (Day 1) to 1 (end of first stomatitis) | 1
  Talking (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Talking (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis) | 1
  Talking (SoC): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Talking (SoC): From 0 (Day 1) to 0 (end of first stomatitis) | 5
  Talking (SoC): From 0 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Talking (SoC): From 0 (Day 1) to 1 (end of first stomatitis) | 1
  Talking (SoC): From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Talking (SoC): From 1 (Day 1) to 0 (end of first stomatitis) | 1
  Talking (SoC): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Talking (SoC): From 2 (Day 1) to 0 (end of first stomatitis) | 1
  Talking (SoC): From 2 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Talking (SoC): From 2 (Day 1) to 1 (end of first stomatitis) | 1
  Talking (SoC): From 3 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Talking (SoC): From 3 (Day 1) to 0 (end of first stomatitis) | 1
  Talking (SoC): From 3 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 13
  Talking (SoC): From 3 (Day 1) to 2 (end of first stomatitis) | 1
  Talking (SoC): From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  Talking (SoC): From missing value (Day 1) to missing value (end of first stomatitis) | 2
  Sleeping (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Sleeping (dexamethasone): From 0 (Day 1) to 0 (end of first stomatitis) | 7
  Sleeping (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Sleeping (dexamethasone): From 1 (Day 1) to 0 (end of first stomatitis) | 1
  Sleeping (dexamethasone): From 2 (Day 1) to 0 (end of stomatitis): number analyzed (Participants) | 11
  Sleeping (dexamethasone): From 2 (Day 1) to 0 (end of stomatitis) | 1
  Sleeping (dexamethasone): From 2 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Sleeping (dexamethasone): From 2 (Day 1) to 1 (end of first stomatitis) | 1
  Sleeping (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Sleeping (dexamethasone): From 2 (Day 1) to 2 (end of first stomatitis) | 1
  Sleeping (SoC): From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Sleeping (SoC): From 0 (Day 1) to 0 (end of first stomatitis) | 5
  Sleeping (SoC): From 0 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 13
  Sleeping (SoC): From 0 (Day 1) to 2 (end of first stomatitis) | 1
  Sleeping (SoC): From 1 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Sleeping (SoC): From 1 (Day 1) to 1 (end of first stomatitis) | 1
  Sleeping (SoC): From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Sleeping (SoC): From 2 (Day 1) to 0 (end of first stomatitis) | 2
  Sleeping (SoC): From 3 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  Sleeping (SoC): From 3 (Day 1) to 0 (end of first stomatitis) | 1
  Sleeping (SoC): From 3 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  Sleeping (SoC): From 3 (Day 1) to 1 (end of first stomatitis) | 1
  Sleeping (SoC): From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  Sleeping (SoC): From missing value (Day 1) to missing value (end of first stomatitis) | 2

20. Secondary Outcome: First-line Treatment (Stomatitis Sub-study): Number of Participants With Shift of Response in OSDQ Score on Mouth Pain Severity at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The fifth item asked the participant to rate their mouth pain severity from 0 (no pain) to 10 (unbearable pain). The mouth pain severity OSDQ scores are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
  Only participants who were randomized in the stomatitis sub-study were included in this analysis.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 24
Participants
  Dexamethasone: From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 0 (Day 1) to 0 (end of first stomatitis) | 1
  Dexamethasone: From 1 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 1 (Day 1) to 2 (end of first stomatitis) | 1
  Dexamethasone: From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 2 (Day 1) to 0 (end of first stomatitis) | 2
  Dexamethasone: From 3 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 3 (Day 1) to 0 (end of first stomatitis) | 2
  Dexamethasone: From 3 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 3 (Day 1) to 1 (end of first stomatitis) | 1
  Dexamethasone: From 3 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 3 (Day 1) to 2 (end of first stomatitis) | 1
  Dexamethasone: From 5 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 5 (Day 1) to 2 (end of first stomatitis) | 1
  Dexamethasone: From 5 (Day 1) to 3 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 5 (Day 1) to 3 (end of first stomatitis) | 1
  Dexamethasone: From 7 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 7 (Day 1) to 1 (end of first stomatitis) | 1
  SoC: From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 1 (Day 1) to 0 (end of first stomatitis) | 1
  SoC: From 1 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 1 (Day 1) to 1 (end of first stomatitis) | 1
  SoC: From 4 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 4 (Day 1) to 1 (end of first stomatitis) | 2
  SoC: From 5 (Day 1) to 5 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 5 (Day 1) to 5 (end of first stomatitis) | 1
  SoC: From 7 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 7 (Day 1) to 0 (end of first stomatitis) | 1
  SoC: From 8 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 8 (Day 1) to 2 (end of first stomatitis) | 1
  SoC: From 8 (Day 1) to 4 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 8 (Day 1) to 4 (end of first stomatitis) | 2
  SoC: From 8 (Day 1) to 6 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 8 (Day 1) to 6 (end of first stomatitis) | 1
  SoC: From 9 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 9 (Day 1) to 0 (end of first stomatitis) | 1
  SoC: From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From missing value (Day 1) to missing value (end of first stomatitis) | 2

21. Secondary Outcome: First-line Treatment (Stomatitis Sub-study): Number of Participants With Shift of Response in OSDQ Score on Mouth Pain Severity Affecting Daily Activities at the End of the First Stomatitis Episode
Description: The OSDQ is a patient self-administered 6-item questionnaire with a 24-hour recall period. Participants completed the questionnaire daily until the resolution of the stomatitis episode. The sixth item asked the participant to rate their mouth pain severity affecting daily activities score from 0 (no effect on daily activities) to 10 (completely prevented from doing daily activities). The mouth pain severity affecting daily activities OSDQ scores are presented as the shift from Day 1 of first stomatitis episode value to the value at the end of the first episode of stomatitis. Day 1 is defined as the first OSDQ questionnaire recorded. End of first stomatitis value is defined as the last OSDQ questionnaire of the first episode of stomatitis. PROs were assessed up to 24 months after last patient's recruitment.
  Only participants who were randomized in the stomatitis sub-study were included in this analysis.
Time Frame: From start date of first stomatitis episode until its resolution, assessed up to 3.8 years
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment)
Number analyzed (Participants) | 24
Participants
  Dexamethasone: From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 0 (Day 1) to 0 (end of first stomatitis) | 5
  Dexamethasone: From 1 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 1 (Day 1) to 0 (end of first stomatitis) | 1
  Dexamethasone: From 2 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 2 (Day 1) to 0 (end of first stomatitis) | 2
  Dexamethasone: From 3 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 3 (Day 1) to 2 (end of first stomatitis) | 1
  Dexamethasone: From 5 (Day 1) to 3 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 5 (Day 1) to 3 (end of first stomatitis) | 1
  Dexamethasone: From 6 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 11
  Dexamethasone: From 6 (Day 1) to 1 (end of first stomatitis) | 1
  SoC: From 0 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 0 (Day 1) to 0 (end of first stomatitis) | 4
  SoC: From 1 (Day 1) to 4 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 1 (Day 1) to 4 (end of first stomatitis) | 1
  SoC: From 2 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 2 (Day 1) to 2 (end of first stomatitis) | 1
  SoC: From 3 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 3 (Day 1) to 0 (end of first stomatitis) | 1
  SoC: From 3 (Day 1) to 1 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 3 (Day 1) to 1 (end of first stomatitis) | 1
  SoC: From 5 (Day 1) to 2 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 5 (Day 1) to 2 (end of first stomatitis) | 1
  SoC: From 5 (Day 1) to 5 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 5 (Day 1) to 5 (end of first stomatitis) | 1
  SoC: From 9 (Day 1) to 0 (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From 9 (Day 1) to 0 (end of first stomatitis) | 1
  SoC: From missing value (Day 1) to missing value (end of first stomatitis): number analyzed (Participants) | 13
  SoC: From missing value (Day 1) to missing value (end of first stomatitis) | 2

22. Secondary Outcome: Number of Participants With Clinical Benfit During Extension Phase
Description: Number of participants with clinical benefit as judged by the investigator during the extension phase. The extension phase for up to 3 years for participants who were continuing to benefit from study treatment following the end of the core study phase (24 months after last patient's recruitment) was added in the amendment 5 (dated 14-Feb-2017). Results are presented by line of treatment
Time Frame: From the end of core phase (upon approval of amendment 5) up to approximately 3 years
Population: For first-line treatment, all participants to whom the first-line treatment was assigned (FAS) For second-line treatment, all participants in the FAS who received at least one dose of second-line study medication (FAS-2L)
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus+Letrozole (First-line Treatment) | Everolimus+Exemestane (Second-line Treatment)
Number analyzed (Participants) | 202 | 53
Participants
  Extension Week 1 | 34 | 6
  Extension Week 12 | 30 | 5
  Extension Week 24 | 28 | 4
  Extension Week 36 | 23 | 3
  Extension Week 48 | 20 | 3
  Extension Week 60 | 18 | 3
  Extension Week 72 | 16 | 3
  Extension Week 84 | 13 | 3
  Extension Week 96 | 12 | 3
  Extension Week 108 | 12 | 3
  Extension Week 120 | 11 | 2
  Extension Week 132 | 10 | 1
  Extension Week 144 | 8 | 1
  Extension End of treatment | 11 | 1

23. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths in first line were collected from first dose of first-line treatment until the date of last administration of the first-line study treatment plus 28 days for participants not entering second-line or the minimum between the date of last administration of the first-line study treatment plus 28 days and the date of first administration of second-line study treatment minus one day for participants entering second line, up to 7.3 years. On-treatment deaths in second line were collected from first dose of second-line treatment to 28 days after the last administration of second-line treatment, up to 5.4 years.
  Post-treatment survival follow-up deaths were collected from day 29 after last dose of study treatment to end of study, up to 7.3 years.
  All deaths refer to the sum of on-treatment deaths and post-treatment deaths.
Time Frame: On-treatment deaths in first line: Up to 7.3 years. On-treatment deaths in second line: Up to 5.4 years. Post-treatment and all deaths: Up to 7.3 years
Population: All participants who received at least one dose of study medication and had at least one post-baseline safety assessment. The safety analysis for the second line was performed on the subset of participants receiving at least one dose of second-line medication.
Measure: Number; unit: Participants
Groups:
- Everolimus + Letrozole/Exemestane (First-line and Second-line Treatment): Participants received everolimus in combination with letrozole as first line treatment. Only participants who had disease progression in the first line setting (core phase) were offered second-line treatment (everolimus in combination with exemestane)
Arm/Group | Everolimus + Letrozole/Exemestane (First-line and Second-line Treatment)
Number analyzed (Participants) | 202
Participants
  On -treatment deaths in first line | 11
  On-treatment deaths in second line: number analyzed (Participants) | 53
  On-treatment deaths in second line | 2
  Post-treatment survival follow-up deaths: number analyzed (Participants) | 125
  Post-treatment survival follow-up deaths | 49
  All deaths | 62

ADVERSE EVENTS:
Time Frame: First-line on-treatment: from the first first-line dose to 28 days post first-line treatment (or 1 day before second-line dose, whichever was earlier, for participants receiving second-line), up to 7.3 years. Second-line on-treatment: from first second-line dose to 28 days post second-line treatment, up to 5.4 years. Post-treatment deaths: from day 29 after final dose to end of study, up to 7.3 years.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up. Deaths in the post treatment survival follow-up are not considered Adverse Events. The total number at risk in the post treatment survival includes patients that entered the post treatment survival follow-up period.
Groups:
- Everolimus+Letrozole (First-line on Treatment): AEs during first-line on-treatment period were collected from the initial first-line dose to 28 days after the last first-line dose, for participants without second-line. For those with second-line treatment, the period lasts until the minimum of 28 days after the last first-line dose or one day before second-line treatment administration.
- Everolimus+Exemestane (Second-line On-treatment): AEs during second-line on-treatment period were collected from first second-line dose to 28 days post second-line treatment
- Everolimus+Letrozole/Exemestane (Post-treatment Survival Follow-up): Deaths collected in the post- treatment survival follow-up period (starting from day 29 after last dose of study treatment). No AEs were collected during this period
Arm/Group | Everolimus+Letrozole (First-line on Treatment) | Everolimus+Exemestane (Second-line On-treatment) | Everolimus+Letrozole/Exemestane (Post-treatment Survival Follow-up)
All-Cause Mortality (participants affected / at risk) | 11/202 | 2/53 | 49/125
Serious Adverse Events (participants affected / at risk) | 72/202 | 8/53 | 0/0
Other Adverse Events (participants affected / at risk) | 202/202 | 43/53 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus+Letrozole (First-line on Treatment) (N=202) | Everolimus+Exemestane (Second-line On-treatment) (N=53) | Everolimus+Letrozole/Exemestane (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 5 | 0 | NA
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0 | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | NA
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | NA
Angina pectoris (Cardiac disorders) | 2 | 0 | NA
Atrial fibrillation (Cardiac disorders) | 4 | 0 | NA
Cardiac failure (Cardiac disorders) | 1 | 0 | NA
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | NA
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | NA
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | NA
Palpitations (Cardiac disorders) | 1 | 0 | NA
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | NA
Vertigo (Ear and labyrinth disorders) | 1 | 0 | NA
Cataract (Eye disorders) | 3 | 0 | NA
Pupils unequal (Eye disorders) | 1 | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | NA
Colitis (Gastrointestinal disorders) | 1 | 0 | NA
Constipation (Gastrointestinal disorders) | 1 | 0 | NA
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | NA
Dysphagia (Gastrointestinal disorders) | 1 | 0 | NA
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | NA
Femoral hernia (Gastrointestinal disorders) | 1 | 0 | NA
Nausea (Gastrointestinal disorders) | 5 | 0 | NA
Odynophagia (Gastrointestinal disorders) | 1 | 0 | NA
Stomatitis (Gastrointestinal disorders) | 1 | 0 | NA
Vomiting (Gastrointestinal disorders) | 4 | 0 | NA
Asthenia (General disorders) | 2 | 0 | NA
Fatigue (General disorders) | 2 | 0 | NA
Non-cardiac chest pain (General disorders) | 1 | 0 | NA
Pyrexia (General disorders) | 2 | 0 | NA
Cholecystitis (Hepatobiliary disorders) | 2 | 0 | NA
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | NA
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | NA
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | NA
Contrast media allergy (Immune system disorders) | 1 | 0 | NA
Abdominal sepsis (Infections and infestations) | 0 | 1 | NA
Appendicitis (Infections and infestations) | 2 | 0 | NA
Cellulitis (Infections and infestations) | 4 | 0 | NA
Clostridium difficile infection (Infections and infestations) | 1 | 0 | NA
Gastroenteritis (Infections and infestations) | 1 | 0 | NA
Hepatitis viral (Infections and infestations) | 0 | 1 | NA
Large intestine infection (Infections and infestations) | 2 | 0 | NA
Paronychia (Infections and infestations) | 1 | 0 | NA
Peritonitis (Infections and infestations) | 1 | 0 | NA
Pneumonia (Infections and infestations) | 9 | 1 | NA
Pneumonia bacterial (Infections and infestations) | 1 | 0 | NA
Pneumonia viral (Infections and infestations) | 1 | 0 | NA
Sepsis (Infections and infestations) | 1 | 0 | NA
Septic shock (Infections and infestations) | 1 | 1 | NA
Soft tissue infection (Infections and infestations) | 1 | 0 | NA
Streptococcal infection (Infections and infestations) | 1 | 0 | NA
Urinary tract infection (Infections and infestations) | 2 | 0 | NA
Vulvitis (Infections and infestations) | 1 | 0 | NA
Accident (Injury, poisoning and procedural complications) | 1 | 0 | NA
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | NA
Snake bite (Injury, poisoning and procedural complications) | 1 | 0 | NA
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | NA
Alanine aminotransferase increased (Investigations) | 0 | 1 | NA
Aspartate aminotransferase increased (Investigations) | 0 | 1 | NA
Blood creatinine increased (Investigations) | 1 | 0 | NA
Ejection fraction decreased (Investigations) | 1 | 0 | NA
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | NA
Weight decreased (Investigations) | 1 | 0 | NA
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | NA
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0 | NA
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 1 | 0 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 5 | 0 | NA
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | NA
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | NA
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | NA
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | NA
Ischaemic stroke (Nervous system disorders) | 1 | 0 | NA
Migraine (Nervous system disorders) | 1 | 0 | NA
Paraesthesia (Nervous system disorders) | 1 | 0 | NA
Syncope (Nervous system disorders) | 1 | 0 | NA
Haematuria (Renal and urinary disorders) | 2 | 0 | NA
Leukocyturia (Renal and urinary disorders) | 1 | 0 | NA
Renal failure (Renal and urinary disorders) | 1 | 1 | NA
Urogenital prolapse (Reproductive system and breast disorders) | 1 | 0 | NA
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | NA
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | NA
Deep vein thrombosis (Vascular disorders) | 1 | 0 | NA
Haematoma (Vascular disorders) | 1 | 0 | NA
Orthostatic hypotension (Vascular disorders) | 1 | 0 | NA
Thrombophlebitis (Vascular disorders) | 1 | 0 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Everolimus+Letrozole (First-line on Treatment) (N=202) | Everolimus+Exemestane (Second-line On-treatment) (N=53) | Everolimus+Letrozole/Exemestane (Post-treatment Survival Follow-up) (N=0)
Anaemia (Blood and lymphatic system disorders) | 71 | 11 | NA
Neutropenia (Blood and lymphatic system disorders) | 15 | 1 | NA
Abdominal pain (Gastrointestinal disorders) | 21 | 4 | NA
Abdominal pain upper (Gastrointestinal disorders) | 15 | 1 | NA
Constipation (Gastrointestinal disorders) | 34 | 1 | NA
Diarrhoea (Gastrointestinal disorders) | 81 | 2 | NA
Dry mouth (Gastrointestinal disorders) | 12 | 0 | NA
Nausea (Gastrointestinal disorders) | 73 | 4 | NA
Oral pain (Gastrointestinal disorders) | 12 | 1 | NA
Stomatitis (Gastrointestinal disorders) | 139 | 10 | NA
Toothache (Gastrointestinal disorders) | 13 | 2 | NA
Vomiting (Gastrointestinal disorders) | 31 | 7 | NA
Asthenia (General disorders) | 32 | 2 | NA
Fatigue (General disorders) | 70 | 5 | NA
Influenza like illness (General disorders) | 7 | 3 | NA
Oedema peripheral (General disorders) | 63 | 6 | NA
Pyrexia (General disorders) | 37 | 3 | NA
Bronchitis (Infections and infestations) | 12 | 4 | NA
Conjunctivitis (Infections and infestations) | 12 | 1 | NA
Gastroenteritis (Infections and infestations) | 11 | 1 | NA
Nasopharyngitis (Infections and infestations) | 29 | 6 | NA
Pneumonia (Infections and infestations) | 27 | 2 | NA
Sinusitis (Infections and infestations) | 14 | 1 | NA
Upper respiratory tract infection (Infections and infestations) | 33 | 4 | NA
Urinary tract infection (Infections and infestations) | 31 | 6 | NA
Alanine aminotransferase increased (Investigations) | 36 | 5 | NA
Aspartate aminotransferase increased (Investigations) | 42 | 5 | NA
Blood cholesterol increased (Investigations) | 42 | 0 | NA
Blood creatine phosphokinase increased (Investigations) | 21 | 7 | NA
Blood creatinine increased (Investigations) | 18 | 3 | NA
Gamma-glutamyltransferase increased (Investigations) | 5 | 3 | NA
Weight decreased (Investigations) | 91 | 15 | NA
White blood cell count decreased (Investigations) | 9 | 3 | NA
Decreased appetite (Metabolism and nutrition disorders) | 64 | 5 | NA
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3 | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 54 | 7 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 59 | 7 | NA
Hyperlipidaemia (Metabolism and nutrition disorders) | 17 | 0 | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 72 | 5 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 32 | 2 | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 14 | 1 | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 59 | 7 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 3 | NA
Bone pain (Musculoskeletal and connective tissue disorders) | 13 | 1 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 4 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 | 2 | NA
Dizziness (Nervous system disorders) | 19 | 1 | NA
Dysgeusia (Nervous system disorders) | 32 | 1 | NA
Headache (Nervous system disorders) | 34 | 4 | NA
Anxiety (Psychiatric disorders) | 16 | 0 | NA
Insomnia (Psychiatric disorders) | 20 | 3 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 70 | 7 | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 48 | 3 | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 36 | 1 | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 15 | 1 | NA
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 12 | 0 | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 | 0 | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 36 | 2 | NA
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 2 | NA
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 4 | 3 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 24 | 1 | NA
Erythema (Skin and subcutaneous tissue disorders) | 15 | 0 | NA
Nail disorder (Skin and subcutaneous tissue disorders) | 12 | 0 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 35 | 1 | NA
Rash (Skin and subcutaneous tissue disorders) | 56 | 0 | NA
Hot flush (Vascular disorders) | 15 | 1 | NA
Hypertension (Vascular disorders) | 50 | 9 | NA
Lymphoedema (Vascular disorders) | 18 | 1 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-02-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT01698918/Prot_000.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/18/NCT01698918/SAP_001.pdf